CLINICAL TRIAL: NCT03474796
Title: Clinical Observation During Anaesthetic Induction: Which Difference Between Novice and Expert ?
Acronym: OCCIA
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Centre Hospitalier Universitaire de Besancon (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: P/2018/361
Record Dates: First submitted 2018-03-09; First posted 2018-03-23 (Actual); Last update posted 2018-03-23 (Actual); Status verified 2018-03

CONDITIONS: Nurse's Role

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Novice (Experimental)
  Interventions: Behavioral: Eye-tracking
- Expert (Experimental)
  Interventions: Behavioral: Eye-tracking

INTERVENTIONS:
Behavioral: Eye-tracking — Visualisation of 4 photographic scenarios (surgical situations), questionnaire, eye-tracking

SUMMARY:
The study aims to show a difference of observation and data integration between novice and expert during anaesthetic induction, in a population of nurse anesthetists.

ELIGIBILITY:
Inclusion Criteria:

* Groupe "novice" : nurse anesthetist students, in 1st or 2nd years at Besançon nursing school OR nurse anesthetists with less than 1 year experience at Besançon University Hospital
* Group "expert" : full-time employed nurse anesthetists, with at least 5 years experience at Besançon University Hospital
* Correct vision with or without correction

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2018-03 (Estimated); Primary Completion 2018-05 (Estimated); Study Completion 2018-06 (Estimated)

PRIMARY OUTCOMES:
Number of eye-fixations on each Region Of Interest (ROI) | Day 1
  Measured with the eye-tracker
Duration of eye-fixation on each ROI | Day 1
  Measured with the eye-tracker

CONTACTS AND LOCATIONS:
Overall Officials: Magali Nicolier, PhD, Principal Investigator — CHU DE BESANCON
Locations (1):
- CHU de Besancon, Besançon, France

IPD SHARING:
Plan to Share IPD: No